CLINICAL TRIAL: NCT05275751
Title: Human Heat Sensation - a Single-group, Randomized, Placebo-controlled, Adaptive, Full-factorial Crossover Trial
Brief Title: Mechanisms of Human Heat Perception - Involvement of TRPA1, TRPV1 and TRPM3
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Heber, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: EK Nr: 1152/2020
Record Dates: First submitted 2022-02-22; First posted 2022-03-11 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Pain
Keywords: Psychophysics; Human physiology; Sensory neuron; TRP channels; Heat perception
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Factorial: There are 4 treatments (TRPV1-, TRPA1-, TRPM3- and chloride channel inhibition). These will be applied in all possible combinations (16). Each healthy volunteer will receive 8 of these 16 combinations in a sequence defined by a Williams square (Hinkelmann, K., and Kempthorne, O. (2005). Design and Analysis of Experiments Vol. 2 - Advanced Experimental Design (Wiley))
  Randomized: Volunteers will be randomly assigned to a pre-specified sequence.
  Placebo-controlled: One of the 16 combinations includes none of the three treatments, i.e., can be regarded as placebo control.
  Adaptive: Due to the complex study design, a priori assumptions about the distribution and correlation of data could not be made reliably. Therefore, after 16 volunteers, the responsible bio-statistician will simulate how much more patients are necessary to detect the a priori defined effect size with the until then observed data
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Hot injection without TRP-channel inhibition (Placebo Comparator): Pain induced by an increasingly hot intradermal injection up to 52°C over 2 minutes.
  Interventions: Drug: Placebo
- Hot injection with TRPA1-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1 is blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor
- Hot injection with TRPV1-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPV1 is blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPV1-inhibitor
- Hot injection with TRPM3-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPM3 is blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPM3-inhibitor
- Hot injection with TRPA1- and TRPV1-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1 and TRPV1 are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPV1-inhibitor
- Hot injection with TRPA1- and TRPM3-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1 and TRPM3 are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPM3-inhibitor
- Hot injection with TRPM3- and TRPV1-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPM3 and TRPV1 are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPV1-inhibitor; Drug: TRPM3-inhibitor
- Hot injection with TRPA1-, TRPV1 and TRPM3-inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1, TRPV1 and TRPM3 are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPV1-inhibitor; Drug: TRPM3-inhibitor
- Hot injection with TRPA1-, TRPM3- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1, TRPM3 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPM3-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPV1-, TRPM3- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPV1, TRPM3 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPV1-inhibitor; Drug: TRPM3-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPA1- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPA1 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPV1- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPV1 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPV1-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPV1-, TRPA1, TRPM3- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPV1, TRPA1, TRPM3 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPV1-inhibitor; Drug: TRPM3-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPM3- and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPM3 and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPM3-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with TRPV1-, TRPA1, and chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while TRPV1, TRPA1, and a chloride channel are blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: TRPA1-inhibitor; Drug: TRPV1-inhibitor; Drug: Chloride-channel inhibitor
- Hot injection with chloride channel inhibition (Experimental): Pain is induced by an increasingly hot intradermal injection up to 52°C over 2 minutes, while a chloride channel is blocked pharmacologically by an antagonist dissolved in the hot fluid (synthetic interstitial fluid). The antagonist(s) have sufficient concentration to reliably block the channel. The total dose is in the range of a microdose trial.
  Interventions: Drug: Chloride-channel inhibitor

INTERVENTIONS:
Drug: TRPA1-inhibitor — Pharmacological inhibition of TRPA1 during intradermal injection of hot synthetic interstitial fluid
  Other Names: Specific antagonist of the TRPA1 channel
  Arms: Hot injection with TRPA1- and TRPM3-inhibition; Hot injection with TRPA1- and TRPV1-inhibition; Hot injection with TRPA1- and chloride channel inhibition; Hot injection with TRPA1-, TRPM3- and chloride channel inhibition; Hot injection with TRPA1-, TRPV1 and TRPM3-inhibition; Hot injection with TRPA1-inhibition; Hot injection with TRPV1-, TRPA1, TRPM3- and chloride channel inhibition; Hot injection with TRPV1-, TRPA1, and chloride channel inhibition
Drug: TRPV1-inhibitor — Pharmacological inhibition of TRPV1 during intradermal injection of hot synthetic interstitial fluid
  Other Names: Specific antagonist of the TRPV1 channel
  Arms: Hot injection with TRPA1- and TRPV1-inhibition; Hot injection with TRPA1-, TRPV1 and TRPM3-inhibition; Hot injection with TRPM3- and TRPV1-inhibition; Hot injection with TRPV1- and chloride channel inhibition; Hot injection with TRPV1-, TRPA1, TRPM3- and chloride channel inhibition; Hot injection with TRPV1-, TRPA1, and chloride channel inhibition; Hot injection with TRPV1-, TRPM3- and chloride channel inhibition; Hot injection with TRPV1-inhibition
Drug: TRPM3-inhibitor — Pharmacological inhibition of TRPM3 during intradermal injection of hot synthetic interstitial fluid
  Other Names: Specific antagonist of the TRPM3 channel
  Arms: Hot injection with TRPA1- and TRPM3-inhibition; Hot injection with TRPA1-, TRPM3- and chloride channel inhibition; Hot injection with TRPA1-, TRPV1 and TRPM3-inhibition; Hot injection with TRPM3- and TRPV1-inhibition; Hot injection with TRPM3- and chloride channel inhibition; Hot injection with TRPM3-inhibition; Hot injection with TRPV1-, TRPA1, TRPM3- and chloride channel inhibition; Hot injection with TRPV1-, TRPM3- and chloride channel inhibition
Drug: Placebo — No pharmacological intervention
  Other Names: No antagonist
  Arms: Hot injection without TRP-channel inhibition
Drug: Chloride-channel inhibitor — Pharmacological inhibition of a chloride channel during intradermal injection of hot synthetic interstitial fluid
  Other Names: Specific inhibitor of a chloride channel
  Arms: Hot injection with TRPA1- and chloride channel inhibition; Hot injection with TRPA1-, TRPM3- and chloride channel inhibition; Hot injection with TRPM3- and chloride channel inhibition; Hot injection with TRPV1- and chloride channel inhibition; Hot injection with TRPV1-, TRPA1, TRPM3- and chloride channel inhibition; Hot injection with TRPV1-, TRPA1, and chloride channel inhibition; Hot injection with TRPV1-, TRPM3- and chloride channel inhibition; Hot injection with chloride channel inhibition

SUMMARY:
Animal studies suggest that the ion channels TRPV1, TRPA1 and TRPM3 are the relevant heat sensors. This study aims to validate these findings in humans.

DETAILED DESCRIPTION:
Surprisingly, it is still not fully understood how humans perceive heat pain. There are several heat-sensitive ion channels whose manipulation in animals resulted in a more or less pronounced phenotype. However, complete blockade of heat sensation in animals has only recently been achieved. In triple knockout mice lacking TRPA1, TRPV1 and TRPM3, it was recently shown that only in the absence of all three receptors heat perception is largely abolished. Although the authors were unable to elucidate the underlying mechanism of this redundancy, the redundancy appears to have evolutionary value for protection against burns. In addition, recent evidence suggests that TRPV1 plays a role as a first-line defense against heat injury, i.e., that it encodes noninjurious heat injury in humans.

The goal of this study is to test whether the redundant functions of TRPV1, TRPA1 and TRPM3 observed in mice with respect to heat perception also apply to humans. More broadly, we want to understand which receptors enable humans to perceive heat pain. The study also aims to test if a chloride channel is involved in heat perception.

Design: Cross-over study with a Williams design group, 16 treatments incl. a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Full legal capacity

To ensure an equal number of each sex in the study population, only volunteers of one sex will be included as soon as the number of subjects with the other sex has reached half of the calculated sample size.

Exclusion Criteria:

* Participant of another study, ongoing or within the last 4 weeks
* Medication intake (except contraception) or drug abuse
* Female subjects: Positive pregnancy test or breastfeeding
* Body temperature above 38°C, diagnostically verified
* Known allergic diseases, in particular asthmatic disorders and skin diseases, known allergic reactions to citrus fruits (but excluding food intolerances).
* Sensory deficit, skin disease or hematoma of unknown origin in physical examination of the test site
* Symptoms of a respiratory tract infection (Covid-19 related criterion)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
HPI(50-52) - Heat pain inhibition in the range between 50°C and 52°C | Through study completion, on average 4 days.
  'Heat pain inhibition between 50 and 52 °C', abbreviated HPI(50-52). A value of 0% would indicate that for a given injection there was no inhibition between 50 and 52 °C, i.e. that the injection was equal to a heated control injection without substance. In contrast, a value of 100% would indicate that there was complete inhibition and the injection was as indistinguishable from the injection at room temperature.
  Of note, pain is rated during the application of the test substances. There are 2 experimental days with injections, separated by a few days, resulting in a time frame of 4 days on average.
  The principle of AUC calculations from pain ratings during injections is described in Heber et al. 2020 (PMID: 32107360 DOI: 0.1097/j.pain.0000000000001848)

SECONDARY OUTCOMES:
HPI - Heat pain inhibition | Through study completion, on average 4 days.
  'Heat pain inhibition between room temperature and 52 °C', abbreviated HPI. A value of 0% would indicate that for a given injection there was no inhibition, i.e. that the injection was equal to a heated control injection without substance. In contrast, a value of 100% would indicate that there was complete inhibition and the injection was as indistinguishable from the injection at room temperature.
  Of note, pain is rated during the application of the test substances. There are 2 experimental days with injections, separated by a few days, resulting in a time frame of 4 days on average.
  The principle of AUC calculations from pain ratings during injections is described in Heber et al. 2020 (PMID: 32107360 DOI: 0.1097/j.pain.0000000000001848)

CONTACTS AND LOCATIONS:
Overall Officials: Michael JM Fischer, Professor MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
All raw data will be shared with other researches upon reasonable request
Supporting Information: Study Protocol, Analytic Code
Time Frame: As soon as the study is published.
Access Criteria: Access will be granted to other researchers as well as clinicians.